CLINICAL TRIAL: NCT02478450
Title: A Phase 1/2a Open-Label Study to Investigate the Safety of the Transplantation (by Injection) of Human Glial Restricted Progenitor Cells (hGRPs; Q-Cells®) Into Subjects With Amyotrophic Lateral Sclerosis (ALS): Assessment of Localized Therapeutic Activity by Blinded Observation and Lateral Transplantation (ALTA-BOLT)
Brief Title: Study to Investigate the Safety of the Transplantation (by Injection) of Human Glial Restricted Progenitor Cells (hGRPs; Q-Cells®) Into Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Q Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QALS-101
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Unilateral lumbar surgical transplantation of Q-Cells dose level 1
  Interventions: Biological: Q-Cells
- Cohort 2 (Experimental): Unilateral cervical surgical transplantation of Q-Cells dose level 1
  Interventions: Biological: Q-Cells
- Cohort 3 (Experimental): Unilateral cervical surgical transplantation of Q-Cells dose level 2
  Interventions: Biological: Q-Cells
- Cohort 4 (Experimental): Unilateral cervical surgical transplantation of Q-Cells dose level 3
  Interventions: Biological: Q-Cells
- Cohort 5 (Experimental): Unilateral cervical surgical transplantation of Q-Cells dose level 4
  Interventions: Biological: Q-Cells
- Cohort 6 (Experimental): Unilateral cervical surgical transplantation of Q-Cells dose level 5
  Interventions: Biological: Q-Cells

INTERVENTIONS:
Biological: Q-Cells — cellular therapeutic comprised of human cells of the glial lineage
  Other Names: glial restricted progenitor cells

SUMMARY:
This study is a non-randomized, open-label, partially blinded, sequential cohort, dose-escalation study designed to obtain preliminary data on the safety, tolerability, and early efficacy of Q-Cells® transplantation in subjects with ALS. Following an initial cohort receiving cell transplants unilaterally in the lumbar spinal cord, subsequent cohorts will receive escalating doses transplanted unilaterally in cervical spinal cord. Subjects and outcome measure assessors will be blinded to side of treatment. The study will be conducted at sites with extensive clinical experience with the care of patients with ALS.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, partially blinded, sequential cohort, dose-escalation study designed to obtain preliminary data on the safety, tolerability, and early efficacy of Q-Cells® transplantation in subjects with ALS. Following an initial cohort receiving cell transplants unilaterally in the lumbar spinal cord, subsequent cohorts will receive escalating doses transplanted unilaterally in cervical spinal cord. Subjects and outcome measure assessors will be blinded to side of treatment. The study will be conducted at sites with extensive clinical experience with the care of patients with ALS.

The study is planned to enroll up to 30 subjects over 24 months. Each subject will receive a single time point administration of Q-Cells®: with 5 or 10 (dependent upon dose level) transplantation foci targeted to the anterior horn in either the lumbar or cervical spinal cord.

The study consists of Screening, Pre-operative/Treatment, and Post-treatment study periods. The study data will be assessed for safety and efficacy after the last subject has completed the 9-month study visit. Following the 9-month study period, subjects who consent will continue to be followed for safety and efficacy long-term in a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to understand the purpose and risks of the study and provide a signed and dated informed consent and authorization to collect and use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Subject lives within reasonable driving distance of study center (approximately 3 hours).
3. Subject has a caregiver willing/able to assist in the transportation and care required by study participation.
4. Subject is 18 - 80 years of age (inclusive) on the first day of the Screening Period.
5. Subject is diagnosed with sporadic or familial ALS within the past 48 months.
6. Subject meets the laboratory-supported probable, clinically probable, or definite criteria for diagnosing ALS according to the World Federation of Neurology El Escorial criteria.
7. Subject has an upright FVC ≥65% of predicted value for age, height, and gender at Screening.
8. Subject has not taken riluzole for at least 30 days prior to the first day of the Screening Period, or has been on a stable dose of riluzole for at least 30 days prior to the first day of the Screening Period (Riluzole-naïve subjects are permitted in the study).
9. Subject is medically able to undergo the study procedures and physically able to adhere to the visit schedule at the time of study entry.
10. Women of childbearing capacity must have a negative pregnancy test during the Screening Period and at the Pre-Operative Visit.
11. Subject must agree to practice effective birth control during study participation.

Exclusion Criteria:

1. Subject in whom causes of neuromuscular weakness other than ALS have not been practically excluded.
2. Subject with a diagnosis of significant cognitive impairment, clinical dementia, or major psychiatric illness including psychosis, bipolar disease, major depression, as determined by the DSM-V.
3. Subject with a diagnosis of other neurodegenerative disease (e.g., Parkinson's disease, Alzheimer's disease).
4. Subject with a diagnosis of any medical condition that impairs nerve or muscle function (e.g., notable peripheral neuropathy, metabolic muscle disease).
5. Subject with a clinically significant history of unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease or other medically significant illness, which, in the opinion of the Investigator, would preclude study participation.
6. Subject with a history of spine surgery or anatomic variation incompatible with route of administration (as determined by neurosurgeon).
7. Subject with severe cervical or lumbar stenosis, cord compression, or cervical or lumbar myelopathy.
8. Subject with abnormal flow voids on the surface of the spinal cord suggestive of arteriovenous malformation (AVM).
9. Subject demonstrating any evidence of CNS malignancy or CNS lesions as defined by imaging studies of the CNS (MRI of brain and spinal cord).
10. Subject having uncontrolled hypertension (Systolic BP>180mmHg and/or Diastolic BP >110mmHg) or having a history of thrombotic events or poorly controlled medical conditions that, in the opinion of the Investigator and/or surgeon, increase risk of surgery.
11. Subject who cannot undergo MRI examination because of the presence of a pacemaker, an implanted defibrillator or certain other implanted electronic or metallic devices, or who have been or might have been exposed to metal fragments, or any reason the subject cannot undergo an MRI routinely for the duration of the trial.
12. Subject with clinically significant abnormal clinical laboratory values, as determined by the Investigator during the Screening Period.
13. Subject who is immune compromised or who has a condition contraindicated to treatment with immunosuppression agents (e.g., tuberculosis, latent infection).
14. Subject with an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value >3.0 times the upper limit of normal or creatinine >1.5 times the upper limit of normal and/or eGFR <50cc/min during the Screening Period.
15. Subject with a history of alcohol or drug abuse or dependence within 1 year of the first day of the Screening Period, per DSM-V criteria.
16. Subject unlikely to comply with study requirements, as determined by Investigator.
17. Subject who has been exposed to any other experimental agent (off-label use or investigational) within 30 days of the first day of the Screening Period. Biologic agents may need additional time for washout and will be evaluated by the Sponsor on a case-by-case basis.
18. Subject who has previously been administered stem cells.
19. Subject with pre-existing anti-human leukocyte antigen (HLA) class I or class II antibodies directed against the Q-Cells®, as determined by panel reactive antibody (PRA) assay during the Screening Period.
20. Subject with an allergy to Q-Cells® or any of its constituents (e.g., chicken eggs), or an allergy to any of the co-administered immunosuppressants or any of their excipients.
21. Subject with any medical condition or using concomitant medication that would contraindicate the use of tacrolimus, mycophenolate mofetil, or prednisone as determined by Investigator.
22. Subject with evidence of deep vein thrombosis (DVT) by venous ultrasound or any previous evidence of DVT.
23. Subject who, in the opinion of the Investigator, has taken or is taking concomitant medications, supplements, or other agents that may interfere with the safety evaluation of Q-Cells® or may affect the course of the subject's ALS progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of human glial restricted progenitor cell transplantation in patients with Amyotrophic Lateral Sclerosis. (adverse events) | 9-month
  Safety will be measured by the number of therapy related adverse events.

SECONDARY OUTCOMES:
Score on the amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 9-month
Quantitative muscle strength values from a hand held dynamometer (HHD) will be tested bilaterally | 9-month
Hand grip (bilateral) values from a grip dynamometer | 9-month
Forced vital capacity (FVC) | 9-month
Maximum sniff nasal inspiratory pressure (SNIP) | 9-month
Electrical Impedance Myography (EIM) values on bilateral upper and lower limbs | 9-month
Pain scores on the Visual Analog Scale (VAS) | 9-month
Score on the ALS Specific Quality of Life Questionnaire - Revised | 9-month
Score on the Ashworth Spasticity Scale | 9-month